CLINICAL TRIAL: NCT00700687
Title: Study Evaluating the Effect on Gastroduodenal Mucosa of PA32540, PA32540 and Celecoxib, and Aspirin With Celecoxib
Acronym: PA32540-109
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: POZEN (Industry)
Responsible Party: Eric Orlemans, POZEN
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PA32540-109
Record Dates: First submitted 2008-06-04; First posted 2008-06-19 (Estimated); Last update posted 2009-01-12 (Estimated); Status verified 2009-01

CONDITIONS: Healthy
Keywords: cardiovascular prophylactic therapy
MeSH Terms: interventions — Celecoxib; Aspirin; Anti-Inflammatory Agents, Non-Steroidal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): PA32540
  Interventions: Drug: PA32540
- 2 (Experimental): PA32540 and celecoxib
  Interventions: Drug: PA32540 and celecoxib
- 3 (Active Comparator): aspirin and celecoxib
  Interventions: Drug: aspirin and [NSAID]

INTERVENTIONS:
Drug: PA32540 — aspirin/omeprazole
  Arms: 1
Drug: PA32540 and celecoxib — aspirin/omeprazole and celecoxib
  Arms: 2
Drug: aspirin and [NSAID] — aspirin and [NSAID]
  Arms: 3

SUMMARY:
We will evaluate the effect on the gastroduodenal mucosa from oral dosing of three different treatments

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or non-pregnant female subjects greater than or equal to 50 years as well as other standard inclusion criteria for a study of this nature

Exclusion Criteria:

* Standard exclusion criteria for a study of this nature

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2008-06; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Lanza scores | entire course of study

SECONDARY OUTCOMES:
safety of three treatments | entrie course of study

CONTACTS AND LOCATIONS:
Locations (1):
- Anaheim, California, United States